CLINICAL TRIAL: NCT03160547
Title: The Effect of Higher Protein Dosing in Critically Ill Patients: A Multicenter Registry-based Randomized Trial
Brief Title: The Effect of Higher Protein Dosing in Critically Ill Patients
Acronym: EFFORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Evaluation Research Unit at Kingston General Hospital (Other)
Responsible Party: Principal Investigator, Daren K. Heyland, Director, Clinical Evaluation Research Unit at Kingston General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: The EFFORT Trial
Record Dates: First submitted 2017-05-17; First posted 2017-05-19 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Critical Illness; Malnutrition
MeSH Terms: conditions — Critical Illness; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Protein/Amino Acid Group (Active Comparator): Patients will receive a usual protein/amino acid dose (≤1.2 g/kg/d)
  Interventions: Other: Usual Protein/Amino Acid Group
- Higher Protein/Amino Acid Group (Active Comparator): Patients will receive a higher protein/amino acid dose (≥2.2 g/kg/d).
  Interventions: Other: Higher Protein/Amino Acid Group

INTERVENTIONS:
Other: Usual Protein/Amino Acid Group — Protein targets will be set using pre-ICU dry actual weight. For patients with BMI >30, ideal body weight based on a BMI of 25 will be used. We will endorse the guidelines for energy targets set forth by ASPEN/SCCM, especially as it pertains to the obese patient.
  Arms: Usual Protein/Amino Acid Group
Other: Higher Protein/Amino Acid Group — Protein targets will be set using pre-ICU dry actual weight. For patients with BMI >30, ideal body weight based on a BMI of 25 will be used. We will endorse the guidelines for energy targets set forth by ASPEN/SCCM, especially as it pertains to the obese patient.
  Arms: Higher Protein/Amino Acid Group

SUMMARY:
The investigator will investigate the effects of higher protein/amino acid dosing (≥2.2 g/kg/d) vs usual protein/amino acid dosing (≤1.2 g/kg/d) on clinical outcomes in nutritionally high risk ill patients.

DETAILED DESCRIPTION:
The EFFORT Study is a multi-center, pragmatic, volunteer-driven, registry-based, randomized, clinical trial of 4000 nutritionally high-risk critically ill patients in the intensive care unit (ICU). We anticipate over 100 sites participating internationally, with each site enrolling a minimum of 30 patients. Patients will be randomized to 1 of 2 treatment groups: a usual prescription (≤1.2 g/kg/d) or a higher prescription (≥2.2 g/kg/d) of protein. Other than the protein amount the patient is randomized to the remainder of care provided to randomized patient will be at the discretion of ICU providers.

In both groups, targets will be achieved through any combination of enteral nutrition (high protein content in high group if available), protein supplements, and parenteral nutrition or amino acids only (as clinically available). The only difference between the 2 groups is the protein targets that are set. Similar efforts should be used in both groups to achieve at least 80% of these targets. The remainder of care provided to eligible patients will be at the discretion of ICU providers.

The investigator has posed two research questions:

Primary Research Question:

In critically ill patients with nutrition 'risk factors', what is the effect of prescribing a higher dose (≥2.2 grams/kg/day) of protein/amino acid administration compared to a usual dose prescribed ≤1.2 gram/kg/day on time to discharge alive from hospital?

Secondary Research Question:

In critically ill patients with nutrition 'risk factors', what is the effect of prescribing a higher dose (≥2.2 grams/kg/day) of protein/amino acid administration compared to patients prescribed ≤1.2 gram/kg/day on 60 day mortality?

The proposed hypothesis:

Compared to receiving usual dose of protein/amino acids, the administration of a higher dose of protein/amino acids (a consequence of having a higher prescription) to nutritionally high-risk critically ill patients will be associated with a quicker rate of recovery and an improved survival.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old
2. Nutritionally 'high-risk' (meeting one of the below criteria)

   1. Low (≤25) or High BMI (≥35)
   2. Moderate to severe malnutrition (as defined by local assessments). We will document the means by which sites are making this determination and capture the elements of the assessment (history of weight loss, history of reduced oral intake, etc.).
   3. Frailty (Clinical Frailty Scale 5 or more from proxy)
   4. Sarcopenia- (SARC-F score of 4 or more from proxy)
   5. From point of screening, projected duration of mechanical ventilation >4 days
3. Requiring mechanical ventilation with actual or expected total duration of mechanical ventilation >48 hours

Exclusion Criteria:

1. >96 continuous hours of mechanical ventilation before screening
2. Expected death or withdrawal of life-sustaining treatments within 7 days from screening
3. Pregnant
4. The responsible clinician feels that the patient either needs low or high protein
5. Patient requires parenteral nutrition only and site does not have products to reach the high protein dose group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1329 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-03 (Actual)

PRIMARY OUTCOMES:
Time to discharge alive from hospital | 60 day
  This is a composite of mortality and length of stay, evaluated up to 60 days post randomization

SECONDARY OUTCOMES:
60-day mortality | 60 day
  Mortality 60 days post randomization

OTHER OUTCOMES:
Nutritional Adequacy | 60 day
  To be evaluated up to 60 days post randomization
Hospital mortality | 60 day
  To be evaluated up to 60 days post randomization
Readmission to ICU and Hospital | 60 day
  To be evaluated up to 60 days post randomization
Duration of Mechanical Ventilation | 60 day
  To be evaluated up to 60 days post randomization
ICU length of stay | 60 day
  To be evaluated up to 60 days post randomization
Hospital length of stay | 60 day
  To be evaluated up to 60 days post randomization

CONTACTS AND LOCATIONS:
Overall Officials: Daren K Heyland, MD, Principal Investigator — Clinical Evaluation Research Unit
Locations (86):
- United States (21):
  - Banner University Medical Center, Phoenix, Arizona
  - Phoenix VA Health Care System, Phoenix, Arizona
  - MemorialCare Long Beach Medical Center, Long Beach, California
  - NorthShore University HealthSystem, Evanston, Illinois
  - SwedishAmercian.Hospital, Rockford, Illinois
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Spectrum Health, Grand Rapids, Michigan
  - Virtua, Marlton, New Jersey
  - Virtua, Mount Holly, New Jersey
  - Virtua, Voorhees Township, New Jersey
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - OU Medical Center, Oklahoma City, Oklahoma
  - Hospital of the University of Pennsylvania - MICU, Philadelphia, Pennsylvania
  - University of Tennessee Medical Center Knoxville, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Virginia Health System, Charlottesville, Virginia
  - Harborview Medical Center, Seattle, Washington
  - Legacy Salmon Creek Medical Center, Vancouver, Washington
  - Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin
- Argentina (2):
  - Hospital Britanico de Buenos Aires, Buenos Aires
  - Sanatorio Allende, Córdoba
- Gold Coast Hospital and Health Service, Gold Coast, Australia
- Brazil (3):
  - Casa de Saude Sao Jose, Rio de Janeiro
  - Hospital e Clinica Sao Goncalo, Rio de Janeiro
  - Hospital Icarai, Rio de Janeiro
- Canada (10):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta, Edmonton, Alberta
  - Abbotsford Regional Hospital, Abbotsford, British Columbia
  - Burnaby Hospital, Burnaby, British Columbia
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Surrey Memorial Hospital, Surrey, British Columbia
  - London Health Sciences Center Hospital, London, Ontario
  - Grey Bruce Health Services, Owen Sound, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - CIUSSS de l'Est-de-l'ile-de-Montreal- Installation Hospital Maisonneuve-Rosemont, Montreal, Quebec
- Greece (2):
  - Agioi Anargiroi Hospital, Athens
  - Evangelismos General Hospital, Athens
- Queen Mary Hospital, Hong Kong, Hong Kong
- Apollo Hospitals Enterprises Limited, Mumbai, India
- Emam Reza Hospital, Mashhad University of Medical Science, Mashhad, Iran
- Japan (2):
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - National Disaster Medical Center, Tokyo, Midori-cho, Tachikawa-shi
- University of Malaya Medical Centre, Kuala Lumpur, Malaysia
- Mexico (4):
  - Hospital San Javier, Guadalajara, Jalisco
  - Hospital Civil Fray Antonio Alcalde, Guadalajara, Jalisco
  - Hospital General Dr. Manuel Gea Gonzalez, Mexico City, Mexico City
  - Hospital Angeles Lomas, México, State of Mexico
- Panama (3):
  - Hospital Regional Rafael Hernandez L. David Chiriqui Css, David, Chiriquí Province
  - Hospital Irma De Lourdes Tzanetatos, Panama City
  - Complejo Hospitalario Dr. Arnulfo Arias Madrid de la Caja de Seguro Social, Panama City
- Hospital Himas San Pablo Caguas, Caguas, Puerto Rico
- King Faisal Specialist Hospital and Research Center, Riyadh, Saudi Arabia
- United Kingdom (32):
  - University Southampton NHS Trust, Southampton, Hampshire
  - Royal Blackburn Hospital, Blackburn
  - North Bristol NHS Trust, Bristol
  - Addenbrooke's Hospital, Cambridge
  - St Richards Hospital, Chichester
  - Northumbria Emergency Care Hospital, Cramlington
  - Royal Infirmary of Edinburgh, Edinburgh
  - Queen Elizabeth Hospital, Gateshead
  - Medway Maritime Hospital, Gillingham
  - Northwick Park hospital, Harrow
  - East Suffolk & North Essex Foundation Trust, Ipswich
  - The Queen Elizabeth Hospital Kings Lynn NHS Trust, Kings Lynn
  - Royal Glamorgan Hospital, Llantrisant
  - Colchester Hospital, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Kings College Hospital Denmark Hill, London
  - Queen Elizabeth Hospital, London
  - Royal Free London NHS Foundation Trust, London
  - University Hospital Lewisham, London
  - Queen Elizabeth the Queen Mother Hospital, Margate
  - Freeman Hospital, Newcastle
  - Aneurin bevan University Health Board, Newport
  - Nottingham University Hospitals NHS Trust, Nottingham
  - The Tunbridge Wells Hospital, Pembury
  - Queen Alexandra, Portsmouth
  - Royal Preston Hospital, Preston
  - Lister Hospital East and North Hertfordshire Trust, Stevenage
  - Royal Stoke Hospital, Stoke-on-Trent
  - Sunderland Royal Hospital, Sunderland
  - Torbay Hospital, Torquay
  - Worthing Hospital, Worthing
  - Yeovil District Hospital NHS Foundation Trust, Yeovil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hoffer LJ, Bistrian BR. Appropriate protein provision in critical illness: a systematic and narrative review. Am J Clin Nutr. 2012 Sep;96(3):591-600. doi: 10.3945/ajcn.111.032078. Epub 2012 Jul 18. PMID 22811443
- [Background] Heyland DK, Cahill N, Day AG. Optimal amount of calories for critically ill patients: depends on how you slice the cake! Crit Care Med. 2011 Dec;39(12):2619-26. doi: 10.1097/CCM.0b013e318226641d. PMID 21705881
- [Background] Jolly SS, Cairns JA, Yusuf S, Meeks B, Pogue J, Rokoss MJ, Kedev S, Thabane L, Stankovic G, Moreno R, Gershlick A, Chowdhary S, Lavi S, Niemela K, Steg PG, Bernat I, Xu Y, Cantor WJ, Overgaard CB, Naber CK, Cheema AN, Welsh RC, Bertrand OF, Avezum A, Bhindi R, Pancholy S, Rao SV, Natarajan MK, ten Berg JM, Shestakovska O, Gao P, Widimsky P, Dzavik V; TOTAL Investigators. Randomized trial of primary PCI with or without routine manual thrombectomy. N Engl J Med. 2015 Apr 9;372(15):1389-98. doi: 10.1056/NEJMoa1415098. Epub 2015 Mar 16. PMID 25853743
- [Background] Fan E, Dowdy DW, Colantuoni E, Mendez-Tellez PA, Sevransky JE, Shanholtz C, Himmelfarb CR, Desai SV, Ciesla N, Herridge MS, Pronovost PJ, Needham DM. Physical complications in acute lung injury survivors: a two-year longitudinal prospective study. Crit Care Med. 2014 Apr;42(4):849-59. doi: 10.1097/CCM.0000000000000040. PMID 24247473
- [Background] De Jonghe B, Sharshar T, Lefaucheur JP, Authier FJ, Durand-Zaleski I, Boussarsar M, Cerf C, Renaud E, Mesrati F, Carlet J, Raphael JC, Outin H, Bastuji-Garin S; Groupe de Reflexion et d'Etude des Neuromyopathies en Reanimation. Paresis acquired in the intensive care unit: a prospective multicenter study. JAMA. 2002 Dec 11;288(22):2859-67. doi: 10.1001/jama.288.22.2859. PMID 12472328
- [Background] Hermans G, Van Mechelen H, Clerckx B, Vanhullebusch T, Mesotten D, Wilmer A, Casaer MP, Meersseman P, Debaveye Y, Van Cromphaut S, Wouters PJ, Gosselink R, Van den Berghe G. Acute outcomes and 1-year mortality of intensive care unit-acquired weakness. A cohort study and propensity-matched analysis. Am J Respir Crit Care Med. 2014 Aug 15;190(4):410-20. doi: 10.1164/rccm.201312-2257OC. PMID 24825371
- [Derived] Tweel LE, Brody R, Samavat H, Day AG, Jiang X, Byham-Gray L, Patel J, Compher C, Heyland DK. Association between protein dose in the early and late acute phases of critical illness and time-to-discharge-alive: A secondary analysis of a randomized clinical trial. JPEN J Parenter Enteral Nutr. 2025 Nov 14. doi: 10.1002/jpen.70033. Online ahead of print. PMID 41236842
- [Derived] Lew CCH, Lee ZY, Day AG, Jiang X, Bear D, Jensen GL, Ng PY, Tweel L, Parillo A, Heyland DK, Compher C. The Association Between Malnutrition and High Protein Treatment on Outcomes in Critically Ill Patients: A Post Hoc Analysis of the EFFORT Protein Randomized Trial. Chest. 2024 Jun;165(6):1380-1391. doi: 10.1016/j.chest.2024.02.008. Epub 2024 Feb 12. PMID 38354904
- [Derived] Haines RW, Prowle JR, Day A, Bear DE, Heyland DK, Puthucheary Z. Association between urea trajectory and protein dose in critically ill adults: a secondary exploratory analysis of the effort protein trial (RE-EFFORT). Crit Care. 2024 Jan 16;28(1):24. doi: 10.1186/s13054-024-04799-1. PMID 38229072
- [Derived] Tweel LE, Compher C, Bear DE, Gutierrez-Castrellon P, Leaver SK, MacEachern K, Ortiz-Reyes L, Pooja L, Leon A, Wedemire C, Lee ZY, Day AG, Heyland DK. A Comparison of High and Usual Protein Dosing in Critically Ill Patients With Obesity: A Post Hoc Analysis of an International, Pragmatic, Single-Blinded, Randomized Clinical Trial. Crit Care Med. 2024 Apr 1;52(4):586-595. doi: 10.1097/CCM.0000000000006117. Epub 2023 Nov 6. PMID 37930244
- [Derived] Stoppe C, Patel JJ, Zarbock A, Lee ZY, Rice TW, Mafrici B, Wehner R, Chan MHM, Lai PCK, MacEachern K, Myrianthefs P, Tsigou E, Ortiz-Reyes L, Jiang X, Day AG, Hasan MS, Meybohm P, Ke L, Heyland DK. The impact of higher protein dosing on outcomes in critically ill patients with acute kidney injury: a post hoc analysis of the EFFORT protein trial. Crit Care. 2023 Oct 18;27(1):399. doi: 10.1186/s13054-023-04663-8. PMID 37853490
- [Derived] Heyland DK, Patel J, Compher C, Rice TW, Bear DE, Lee ZY, Gonzalez VC, O'Reilly K, Regala R, Wedemire C, Ibarra-Estrada M, Stoppe C, Ortiz-Reyes L, Jiang X, Day AG; EFFORT Protein Trial team. The effect of higher protein dosing in critically ill patients with high nutritional risk (EFFORT Protein): an international, multicentre, pragmatic, registry-based randomised trial. Lancet. 2023 Feb 18;401(10376):568-576. doi: 10.1016/S0140-6736(22)02469-2. Epub 2023 Jan 25. PMID 36708732
- [Derived] Hill A, Heyland DK, Elke G, Schaller SJ, Stocker R, Haberthur C, von Loeffelholz C, Suchner U, Puthucheary ZA, Bear DE, Ney J, Clasen KC, Meybohm P, Lindau S, Laurentius T, Stoppe C. Meeting nutritional targets of critically ill patients by combined enteral and parenteral nutrition: review and rationale for the EFFORTcombo trial. Nutr Res Rev. 2020 Dec;33(2):312-320. doi: 10.1017/S0954422420000165. Epub 2020 Jul 16. PMID 32669140

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2017-10-01): https://cdn.clinicaltrials.gov/large-docs/47/NCT03160547/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2022-03-09): https://cdn.clinicaltrials.gov/large-docs/47/NCT03160547/SAP_001.pdf